CLINICAL TRIAL: NCT01878448
Title: Phase 2 Study of Anlotinib in Advanced Soft Tissue Sarcoma
Brief Title: A Phase II Study of Anlotinib in STS Patients
Acronym: ALTN/STS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-02-II
Record Dates: First submitted 2013-05-30; First posted 2013-06-17 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — anlotinib

ARMS (1):
- Anlotinib (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib

SUMMARY:
Anlotibib (ALTN) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd.

ALTN is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2 and VEGFR3. It has the obvious resistance to new angiogenesis. The protocol is to explore ALTN for the effectiveness of advanced soft tissue sarcoma and security.

ELIGIBILITY:
Inclusion Criteria:

* 1.Faild in introditional treatmeat, Mainly includes:MFH/liposarcoma/leiomyosarcoma/SS and others(MPNST/Fibrosarcoma/CCS/ASPS/AS/ES; 2.Receiveed at least one chemotherapy regimens treatment; 3.18-70years, ECOG:0-2,Expected survival period >3 months; 4.HB≥100g/L,ANC(Absolute Neutrophil Count) ≥1.5×109/L；PLT

  * 80×109/L ,BIL/Cr in normal range,ALT/AST(aspartate aminotransferase )≤1.5*ULN(for hepatic metastases,ALT/AST(aspartate aminotransferase )≤5*ULN) ;TG≤ 3.0mmol/L，cholesterol≤7.75mmol/L; LVEF
  * LLN. 5.Used contraceptive during the study and after 6 months; 6.Volunteer.

Exclusion Criteria:

* 1. Received vascular endothelial growth inhibitor type of targeted therapy; 2.With the second cancer; 3.Participated in other clinical trials in four weeks; 4.Received in other radiotherapy or chemotherapy treatment in four weeks; 5.AE>1 6.Has influence of oral drugs; 7.Brain metastases, spinal cord compression, cancerous meningitis; 8.Any serious or failed to control the disease 9.Artery/venous thrombotic; 10.Coagulant function abnormality; 11.Arteriovenous thrombosis event; 12.Hitory of psychiatric drugs abuse or a mental disorder; 13.Immunodeficiency history; 14.Concomitant diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-04; Primary Completion 2015-10 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
tumor size | each 42 days up to 48 months
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule by enhanced CT scan every two cycles. Refer to recist 1.1.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | each 21 days up to 48 months
  blood examination, urine examination, stool examination, blood biochemical (ALT, AST, TB(total bilirubin), DB, BUN, Cr, blood electrolyte), electrocardiogram (ecg), thyroid function, the function of blood coagulation, etc

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The 1st affiliated hospital of bengbu medical college, Bengbu, An'hui
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Province Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Meidical University, Fuzhou, Fujian
  - Gansu Province Tumor Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi medical university affiliated tumor hospital, Nanning, Guangxi
  - Harbin medical university affiliated tumor hospital, Harbin, Heilongjiang
  - Liaoning Province Tumor Hospital, Shenyang, Liaoning
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality